CLINICAL TRIAL: NCT01616537
Title: Evaluation of Patient Satisfaction With and Acceptance of Their Totally-implanted Central Venous Catheter: Confirmatory Validation of QASICC Questionnaire
Brief Title: Evaluation of Patient Satisfaction With and Acceptance of Their Totally-implanted Central Venous Catheter
Acronym: QASICC-EVA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011-A01063-38
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2013-02

CONDITIONS: Malignant Mast Cell Tumors; Solid Organ Sites
Keywords: solid tumors; hematological malignancy
MeSH Terms: conditions — Mast-Cell Sarcoma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: QUALITY OF LIFE QUESTIONNAIRE — QASICC AND EORTC QLQ-C30 ADMINISTRATION 30 DAYS AFTER CVC IMPLANTATION
  Other Names: QASICC; EORTC QLQ-C30

SUMMARY:
Background Patient satisfaction with or acceptance of care assessment is increasingly taken into account in oncology. Most cancer and other critically-ill patients require a totally-implanted Central Venous Catheter (CVC) for their treatment consisting of a reservoir connected to a central venous catheter, which may or may not be valved. It is impossible to estimate the number of CVC used in oncology. However, some authors claim that, in 2005, over 7 million CVCs were placed in the United States in both chronic and acute care. Although many patients fitted with a CVC are able to undertake activities which are hindered with other external vascular access devices, they are often physically or psychologically anxious about their device. To our knowledge, no validated questionnaire measuring patient acceptance of and satisfaction with their CVC has been reported in the literature. Based on these observations, the aim of our study was to develop and to validate a French-language questionnaire dubbed QASICC (Questionnaire for Acceptance of and Satisfaction with Implanted Central Venous Catheter) assessing patient satisfaction with and acceptance of their CVC. QASICC is designed as a multi-dimensional, self-administered questionnaire comprising approximately 30 items related to the use, appearance and pros and cons of the device as well as quality of life as perceived by patients using one for treatment.

Objective The purpose of the study is to validate a French-language self-administered questionnaire (QASICC) designed to evaluate patients' satisfaction and acceptance concerning their totally-implanted central venous catheter: confirmatory validation of questionnaire psychometric properties.

Study Design This is a prospective, multicenter, open study.

Primary Outcome Measures:

Questionnaire's 27 items tested on 990 patients to confirm QASICC internal structure:

* Items quality
* Dimensional structure
* Dimensional consistence
* Measure accuracy
* Measure reliability
* Sensitivity to change

DETAILED DESCRIPTION:
QASICC Questionnaire The QASICC questionnaire included 27 questions (Q) assessing seven dimensions: pain during placement or use (Q1, Q2), contribution to the comfort of the treatment (Q3, Q4, Q7, Q10, Q12), esthetics and privacy (Q5, Q6, Q8, Q11, Q17, Q19), the impact on professional activities, social and sports (Q9, Q13, Q14, Q18, Q20), the impact on daily activities (Q15, Q16, Q21, Q22 ), local discomfort (Q23, Q24, Q25, Q26) and overall satisfaction (Q27). The device-related answers were of two types: Likert or visual analogue scale. Four types of Likert response were available: "no", "low," "moderate," "significant,"/"never," "sometimes," "often," "always "/" very easy "," easy "," difficult "," very difficult "/" not at all "," somewhat "," a lot "," extremely ". These questions are scored 0, 33, 67, 100, respectively, when the scores are correlated with symptoms, or 100, 67, 33, 0 when the scores are inversely correlated with symptoms. Visual analog scales (VAS) have a length of 100 mm. The score represents the number of mm measured on the scale. A mean score of acceptance and satisfaction can be calculated on a scale of 0 to 100 for all seven dimensions using the following formula: {(100-score DO) + CO + score (score ES-100) + (100-PR score) + (100-ES score) + (score 100-IN) + SA score} / 7. The higher the overall score, the greater the acceptance and satisfaction

The questionnaire is administered to the patient 30 days (+/-7 days) after CVC implantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patient who benefited or will benefit from the implantation of a CVC
* Solid tumor or hematologic malignancy
* WHO Performance Status 0-2

Exclusion Criteria:

* Any severe psychopathological disorder preventing completion of the questionnaire or invalidating questionnaire's measures
* Severe depressive state
* Non malignant pathology
* Inability to respond to questionnaires
* Patient not speaking fluent French
* Patient unable to consent
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
QASICC questionnaire's 27 items tested on 990 patients to confirm the internal structure | 30 days (+/- 7 days) after CVC implantation
  * Items quality
  * Dimensional structure
  * Dimensional consistence
  * Measure accuracy
  * Measure reliability
  * Sensitivity to change

SECONDARY OUTCOMES:
Questionnaire's 27 items tested on 990 patients to confirm QASICC external structure: convergent-divergent validity compared to EORTC-QLQC30 questionnaire. | 30 days (+/-7 days) after CVC implantation
  convergent-divergent validity of the QASICC questionnaire compared to EORTC-QLQC30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: PIERRE YVES MARCY, MD, Principal Investigator — Centre Antoine Lacassagne
Locations (10):
- France (10):
  - Centre Paul Papin - Ico, Angers
  - Centre Francois Baclesse, Caen
  - Chu La Timone, Marseille
  - Chu de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Jean Godinot, Reims
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy